CLINICAL TRIAL: NCT01184768
Title: HBA1c and Diagnosis of Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: University of Tromso (Other)
Responsible Party: Rolf Jorde, University of Tromsø
Other Study IDs: UIT-ENDO-2010-2
Record Dates: First submitted 2010-08-11; First posted 2010-08-19 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; HbA1c; vitamin D; diagnosis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- participants in the 6th tromsø study

SUMMARY:
Following the 6th Tromso study subjects with HbA1c > 5.7 plus a subsample of subjects with lower hba1c values will be invited to an oral glucose tolerance test to see the predictive value of HBA1c in the diagnosis of type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* participated in the 6 Tromso study

Exclusion Criteria:

* type 2 diabetes

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: random sample of subjects living in Tromso and who participated in the 6 th Tromsø study
Sampling Method: Non-Probability Sample
Enrollment: 3509 (Actual)
Dates: Start 2008-01; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Number of subjects with new diagnosis of type 2 diabetes | Up to 2 years after participation in the 6th Tromso study

SECONDARY OUTCOMES:
Number of subjects with new diagnosis of impaired glucose tolerance | Up to 2 years after participation in the 6th Tromso study
Number of subjects with new diagnosis of impaired fasting glucose | Up to 2 years after participation in the 6th Tromso study
Effect of vitamin D status on glucose tolerance | Up to 2 years after participation in the 6th Tromso study

CONTACTS AND LOCATIONS:
Overall Officials: rolf jorde, md, Principal Investigator — University of Tromso
Locations (1):
- University Hospital of North Norway, Tromsø, Tromsø, Norway